CLINICAL TRIAL: NCT05784766
Title: Screening for Atrial Fibrillation in Patients With Cancer: A Pilot Randomized Controlled Clinical Trial
Acronym: SARIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15595
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Screen group (Active Comparator): Patients randomized to screening will undergo a 30-second ECG using the Kardia Mobile device (AliveCor Inc, Cupertino, CA) paired with an iPad (Apple, Cupertino, CA). If the mobile ECG shows possible AF or unclassified, then patients will undergo a 12-lead standard ECG during the same visit, read by a cardiologist, to verify the correct diagnosis.
  Interventions: Diagnostic Test: 30-second ECG using the Kardia Mobile
- Usual Care (Active Comparator): For patients in the usual care arm, medical record review will be done at end of study to assess for the newly diagnosed AF during the study period.
  Interventions: Other: routine care

INTERVENTIONS:
Diagnostic Test: 30-second ECG using the Kardia Mobile — 30-second ECG using the Kardia Mobile
  Arms: Screen group
Other: routine care — medical review
  Arms: Usual Care

SUMMARY:
Patients with cancer have a higher incidence of AF but despite the higher incidence of AF in the cancer population, there are no randomized controlled trials (RCTs) for AF screening in this population. RCTs of AF screening in the general population have shown that screening can effectively detect AF earlier, and helps to identify candidates for appropriate anticoagulation that may lead to improvement in clinical outcomes.

DETAILED DESCRIPTION:
The Investigators will conduct an open label, prospective, pilot RCT. After informed consent, patients will be randomized 1:1 into screening or usual care. Screening will be done at a single time point. Patients randomized to screening will undergo a 30-second ECG using the Kardia Mobile device (AliveCor Inc, Cupertino, CA) paired with an iPad (Apple, Cupertino, CA). Patients randomized to usual care will not receive a screening ECG. Primary outcome will be detection of newly diagnosed AF by screening vs usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age ≥65 with a current diagnosis or history of cancer.
2. Patients currently undergoing or history of chemotherapy, radiotherapy or cancer related surgeries will be included.
3. The age is restricted to ≥65 years because prevalence of AF is extremely low. .

Exclusion Criteria:

1. Known history of atrial fibrillation.
2. Non-English-speaking participants will not be enrolled

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The Investigators will compare the incidence of newly diagnosed AF identified by screening versus usual care | 6 MONTHS
  To compare the incidence of newly diagnosed AF with point-of-care screening using a mobile, single-lead ECG versus usual care, in patients with a diagnosis of solid cancer. In this open-label, prospective pilot RCT, patients (n=480) with AF and solid cancer presenting for an outpatient visit will be randomized 1:1 to screening versus usual care. A 30-second screening ECG will be done using the Kardia Mobile device (AliveCor Inc, Cupertino, CA) paired with an iPad. The Investigators will compare the incidence of newly diagnosed AF identified by screening versus usual care.

SECONDARY OUTCOMES:
To determine the effect of screening-detected AF on initiation of anticoagulation. | 6 MONTHS
  To determine the effect of screening-detected AF on initiation of anticoagulation. Patients diagnosed with AF through screening will be referred to their primary care physician for initiation of anticoagulation based on their CHA2DS2VASc score.The Investigators will conduct chart review at the end of study to compare the proportion of patients appropriately initiated on anticoagulation between screening versus usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Zain Asad, MD, Principal Investigator — OU Health
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States